CLINICAL TRIAL: NCT00943774
Title: Blood Pressure Variability, Baroreflex Sensitivity, and Cardiovascular Responses to Sympathoexcitation in Healthy Normotensive Humans
Brief Title: High Resolution Phenotyping in Healthy Humans
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John Eisenach, PI, Mayo Clinic
Other Study IDs: 05-004352; R01HL089331 (NIH); NS-32352
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Pressor Response; Baroreflex Sensitivity; Blood Pressure Variability; Heart Rate Variability; Arterial Catecholamines
Keywords: Physiology; Phenotype; Genetics; Genomics; Stress; Baroreflex; Blood Pressure; Arterial stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, white cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All subjects: All subject participants
  Interventions: Other: Physiological maneuvers

INTERVENTIONS:
Other: Physiological maneuvers — These healthy subjects undergo physiological testing, which includes aortic augmentation index, pulse wave velocity, orthostatic stress, baroreflex sensitivity (modified Oxford protocol), mental stress, cold pressor test, isometric handgrip, heart rate variability, 24-hour ambulatory blood pressure monitoring.

SUMMARY:
Baroreflex sensitivity is integral to blood pressure regulation, and varies among healthy, normotensive individuals. A reduced compensatory ability of baroreflex buffering in patients with carotid denervation results in blood pressure variability and an elevated blood pressure response to mental stress. Furthermore, 24-hour ambulatory blood pressure variability may also be a significant and independent risk determinant of cardiovascular disease. It remains unknown whether the degree of baroreflex sensitivity and ambulatory blood pressure variability are predictive of the pressor response to sympathoexcitatory stress in healthy humans. In this study the investigators propose a comprehensive evaluation of the relationships among the pressor and forearm vasodilator response to sympathoexcitation, ambulatory blood pressure variability, and baroreflex sensitivity in healthy normotensive subjects. Ultimately this study will provide preliminary data and protocol development for large-scale high resolution phenotyping in population-based trials aimed at determining the functional relevance of candidate gene variation in intermediate physiological traits pertinent to the pathogenesis of hypertension and cardiovascular disease.

DETAILED DESCRIPTION:
Growing evidence suggests an association of environmental stress with the development of hypertension and there is strong evidence in normotensive subjects that a greater pressor response to sympathoexcitatory stress is a harbinger of future hypertension. Pharmacological studies have shown that individuals with HTN have a blunted baroreflex sensitivity, and display a greater increase in blood pressure during administration of an alpha-agonist. Furthermore, exaggerated 24-hour ambulatory blood pressure variability (BPV) is proposed to be a risk factor for the development of cardiovascular disease. Finally, Beta-2 adrenergic receptor-mediated forearm vasodilator responses to mental stress are blunted in Caucasian subjects at increased risk for hypertension, in African Americans, and in mild hypertension. We postulate that a relationship exists between these variables, even in normotensive healthy individuals. We also believe that signs of subclinical metabolic dysfunction exist in healthy individuals and that they may either contribute to or be affected by BPV. There is also evidence the prematurity at birth and low birth weight are associated with hypertension. Finally, arterial stiffness may also be related to blood pressure variability and the pressor response. Therefore the specific aims of this study are:

1. To examine the relationship between 24-hour ambulatory BPV and baroreflex sensitivity. By measuring the baroreflex control of heart rate during sequential boluses of nitroprusside and phenylephrine, we hypothesize that baroreflex sensitivity will be inversely related to the degree of 24-hour BPV.
2. To examine the relationship between 24-hour ambulatory BPV and the pressor response to four sympathoexcitatory maneuvers: head-up tilt testing, mental stress, cold pressor test, and isometric handgrip to fatigue. We hypothesize that greater BPV will predict the pressor response to stress.
3. To examine the relationship between baroreflex sensitivity and the pressor response/forearm vasodilator response to the three sympathoexcitatory maneuvers. We hypothesize that individuals with higher baroreflex sensitivity will have a lower pressor response and a lower forearm vasodilator response to sympathoexcitatory stress.
4. To draw a venous blood sample for future screening of genetic polymorphisms of interest, which may include nitric oxide synthase (NOS), alpha-adrenergic and beta-adrenergic receptor polymorphisms. We hypothesize that genetic variation in these key regulatory systems might explain some of the differences in baroreflex sensitivity, BPV, the pressor response and forearm vasodilator response to sympathoexcitation.
5. To examine the relationship between 24-hour ambulatory BPV and the pressor response to sympathoexcitatory maneuvers and insulin resistance, dyslipidemia, and body fat distribution. We hypothesize that greater BPV will be associated with insulin resistance, dyslipidemia, and increase waist-hip ratio.
6. To examine the relationship between 24-hour ambulatory BPV and arterial stiffness using measurements of pulse wave velocity. We hypothesize that greater BPV will be associated with increased pulse wave velocity, an index of arterial stiffness.
7. To examine the relationship between 24-hour ambulatory BPV and the pressor response to sympathoexcitatory maneuvers with birth weight and post-conceptual age at birth. We will ask each subject to provide this data based on their birth certificate and/or knowledge of their medical history.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18-40
* Non-pregnant women age 18-50

Exclusion Criteria:

* Any medical conditions affecting the cardiovascular system
* Any prescribed chronic medications (except contraceptives)
* Extremes of fitness (not totally sedentary, not highly exercise-trained)
* BMI greater than 28

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Southeast Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Response to Sympathoexcitation | On day of study

SECONDARY OUTCOMES:
Baroreflex Sensitivity | On day of study

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Ramirez-Marrero FA, Charkoudian N, Hart EC, Schroeder D, Zhong L, Eisenach JH, Joyner MJ. Cardiovascular dynamics in healthy subjects with differing heart rate responses to tilt. J Appl Physiol (1985). 2008 Nov;105(5):1448-53. doi: 10.1152/japplphysiol.90796.2008. Epub 2008 Aug 28. PMID 18756006
- [Result] Ramirez-Marrero FA, Charkoudian N, Zhong L, Hesse C, Eisenach JH. Balance between sympathetic response to head-up tilt and cardiac vagal factors in healthy humans. Clin Auton Res. 2007 Aug;17(4):227-30. doi: 10.1007/s10286-007-0427-y. Epub 2007 Aug 23. PMID 17717719
- [Result] Hesse C, Charkoudian N, Liu Z, Joyner MJ, Eisenach JH. Baroreflex sensitivity inversely correlates with ambulatory blood pressure in healthy normotensive humans. Hypertension. 2007 Jul;50(1):41-6. doi: 10.1161/HYPERTENSIONAHA.107.090308. Epub 2007 May 14. PMID 17502489